CLINICAL TRIAL: NCT07095192
Title: Scaling Up Point-of-Care Hepatitis C Testing and Treatment in Canada: A Multilevel Implementation Science Study of Clinical Processes, Barriers, Facilitators and Implementation Strategies
Brief Title: Scaling Up Point-of-Care Hepatitis C Testing and Treatment in Canada
Acronym: SCALE POCT
Status: Recruiting | Type: Observational
Sponsor: McGill University (Other)
Collaborators: The University of New South Wales (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Jewish General Hospital (Other); University of British Columbia (Other); British Columbia Centre for Disease Control (Other Government); University of Toronto (Other); York University (Other); Ottawa Hospital Research Institute (Other); University of Ottawa (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Lady Davis Institute (Other); International Network on Health and Hepatitis in Substance Users (Unknown); Public Health Agency of Canada (PHAC) (Other Government); Canadian Association of People who Use Drugs (Unknown); Action Hepatitis Canada (Unknown); Canadian Liver Foundation (Unknown); CATIE (Unknown); Canadian Network on Hepatitis C (Unknown)
Responsible Party: Principal Investigator, Guillaume Fontaine, Assistant Professor, McGill University
Other Study IDs: 24-12-038; PJT- 517467 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-07-03; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: HCV; HEPATITIS C VIRUS CHRONIC INFECTION
Keywords: HCV; Hepatitis C Virus Chronic Infection; Rapid point-of-care testing; Implementation science; Knowledge translation; Marginalized populations; Infectious diseases; Barriers and facilitators; Implementation strategies
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Consumers: Individuals aged ≥18 years who have a risk factor for HCV acquisition or are attending a site that provides services to people with an HCV acquisition risk
  Interventions: Other: Preimplementation of HCV Point of care testing
- Provider and manager: Participants must be currently employed at one of the research sites and involved in or supervising the delivery of HCV-related services.
  Interventions: Other: Preimplementation of HCV Point of care testing
- Decision-maker: Participants must hold a position in local, provincial, or national government, health authority or another organization that influences HCV testing and treatment policies and be able to provide insights into the strategic planning and funding for HCV care.
  Interventions: Other: Preimplementation of HCV Point of care testing
- Laboratory and quality assurance stakeholder: Participants must hold a role in laboratory services, quality assurance, or regulatory oversight of point-of-care testing at the provincial, national, or organizational level.
  Interventions: Other: Preimplementation of HCV Point of care testing

INTERVENTIONS:
Other: Preimplementation of HCV Point of care testing — Exploring the pre-implementation of HCV Point of care antibody and RNA tests

SUMMARY:
The SCALE-POCT study is a national initiative designed to provide robust evidence for scaling up point-of-care hepatitis C testing for key populations. The study seeks to map current hepatitis C clinical processes, identify barriers and facilitators to implementation, and co-design practical tools and strategies in partnership with stakeholders.

A major obstacle to hepatitis C elimination and increasing treatment uptake is the current multi-step diagnostic process, which leads to loss to follow-up and treatment delays, particularly among high-risk groups such as people who inject drugs. Point of-care hepatitis C antibody tests (results: 5-20 mins) and RNA tests (results: 60 mins), could enable single-visit diagnosis, reducing loss to follow-up. However, integrating these tests into key settings presents challenges. The overarching goal of this study is to generate evidence to inform the scale-up point-of-care hepatitis C testing and treatment in key settings in Canada. This study is observational in nature and does not involve the direct implementation of point-of-care hepatitis C testing. Instead, it aims to understand the contextual, procedural, and operational factors that would support its successful adoption and sustainability. By examining existing care models and engaging with key stakeholders, the study seeks to build a foundation for future implementation efforts. Specific objectives include:

1. Map current hepatitis C care processes and explore how point-of-care testing could fit into these models;
2. Identify barriers and facilitators to implementing point-of-care hepatitis C testing across settings and provinces;
3. Co-design tools and strategies (such as training guides, standard procedures) to support point-of-care testing;
4. Assess feasibility, acceptability, and costs of the co-designed tools and strategies.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a major public health threat in Canada (~204,000 people living with HCV in 2019. HCV therapies with cure >95% are one of the greatest medical advances in decades and have led the WHO to set a goal to eliminate HCV by 2030. In Canada, achieving elimination will require significant increases in diagnoses and treatment . A major barrier to increasing uptake of HCV testing/treatment is that the current diagnostic pathway requires multiple visits (an HCV antibody test to confirm exposure, an HCV RNA test to confirm current infection, and one or more assessments to start treatment) leading to loss to follow-up and delays in treatment. This is amplified in populations with the highest HCV burden, including people who inject drugs (85% of new infections; 46.1% prevalence) and those in prison (10.7% prevalence). People who inject drugs face barriers to accessing HCV care including stigma/discrimination (leading to avoidance of healthcare), inadequate health service access, and poor venous access (making blood collection for testing difficult), whereas people in prison are often released prior to their antibody or RNA result (2, 4, 5). There is an urgent need to leverage innovations to streamline the diagnostic pathway and enhance access to testing/treatment.

The introduction of finger-stick tests capable of detecting HCV antibodies (results: 5-20 minutes) and HCV RNA (results: 60 minutes) at the point-of-care has revolutionized the clinical approach to HCV. These point-of-care tests enable diagnosis and treatment in a single visit, increase testing acceptability, and reduce loss to follow-up. Research by our team has demonstrated excellent technical accuracy and clinical utility of these tests, with pilot studies showing high treatment uptake compared to standard diagnostic approaches, informing recommendation in the 2022 WHO Guidelines and their forthcoming approval by Health Canada. Our team has developed a program for the implementation of point-of-care HCV testing in Australia, resulting in rapid national scale-up across 90 sites, with 20,000 tests and >1,500 people treated (79% treatment uptake; 93% in prisons).

Point-of-care HCV antibody and RNA testing is a 'game-changing' solution to address a critical gap in care and increase equity in healthcare access, particularly for marginalized groups, as we seek to achieve our national elimination targets. The impact of point-of-care testing will be greatest in high HCV prevalence settings (those caring for people who inject drugs), such as needle and syringe programs, drug treatment, prisons, and outreach settings. However, implementation challenges persist, including quality assurance and integration of point-of-care tests into diverse laboratory/public health surveillance frameworks. A systematic, implementation science-based approach is essential to comprehensively identify factors that will limit or enable point-of-care HCV testing within the Canadian context. This is critical for developing specific implementation strategies that address barriers and amplify facilitators to point-of-care testing, and informing changes to health service delivery, guidelines, and provincial and national strategies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥18 years who have a risk factor for HCV acquisition or are attending a site that provides services to people with an HCV acquisition risk.
* Service providers and managers who are currently employed at a site providing HCV-related services, involved in or supervising the delivery of HCV-related services.
* Policymaker must hold a position in local, provincial, or national government or a health authority that influences HCV testing/treatment policies and be able to provide insights into the strategic planning and funding for HCV care.
* Laboratory and quality assurance stakeholders must hold a role in laboratory services, quality assurance, or regulatory oversight of point-of-care testing at the provincial, national, or organizational level.

Exclusion Criteria:

* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults at risk of HCV (current/past injecting drug use, current/previous incarceration, HIV, having a tattoo/piercing in an unregulated environment).
  Providers (e.g., physicians, nurses, harm reduction workers, street workers) and managers who work with those at risk of HCV, involved in or supervising the delivery of HCV-related services.
  Decision-makers: People who hold a position in local, provincial, or national government, health authority, or another organization that influences HCV testing and treatment policies and be able to provide insights into the strategic planning and funding for HCV care.
  Laboratory and quality assurance stakeholders: People who provide laboratory services, quality assurance, or regulatory oversight of point-of-care testing at the provincial, national, or organizational level.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-06-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Measure Barriers and facilitators based on the CFIR Constructs | 1 year
  Using the ERIC Taxonomy and the CFIR-ERIC Matching Tool, we will link identified barriers and facilitators to evidence-based implementation strategies. The ERIC Taxonomy includes 73 strategies across 9 clusters, such as training stakeholders, supporting clinicians, engaging consumers, and changing infrastructure. This step will produce a matrix that maps each barrier and facilitator to one or more relevant strategies.
Acceptability and Feasibility of Point-of-Care Testing Strategies (Provider/Manager Survey, Section 2) | 1 year
  The questionnaire adapts the Intervention Appropriateness Measure (IAM) and Feasibility of Intervention Measure (FIM) to assess acceptability and feasibility. Each strategy is evaluated with 8 Likert-scale questions (1-5). Data will be aggregated as mean scores, with higher scores (minimum score: 8, maximum score: 40) indicating greater perceived acceptability/feasibility.
Acceptability and Feasibility of Point-of-Care Testing Strategies (Provider/Manager Survey, Section 3) | 1 year
  The questionnaire adapts the Organizational Readiness for Implementing Change (ORIC) tool to assess feasibility by evaluating if the organization has the commitment and confidence in its ability to implement change. Feasability is assessed through with 12 Likert-scale questions (1-5, minimum score: 12, maximum score: 60)
Sustainability of Point-of-Care Testing Strategies using the Time-driven activity-based costing (TDABC) | 1 year
  Time-driven activity-based costing methodology will guide assessment of costs incurred by health resource use during the patient care cycle to determine the sustainability of the point-of-care testing. This will be done by: 1) determining the frequency, capacity, and average duration of each implementation action by actors, as well as actors' total time spent on each action; 2) determine the price per hour of each actor; 3) determine non-personnel, fixed resources, and their associated expenses; 4) creation and use of a TDABC resource costing matrix to blueprint site-specific implementation processes and calculate total costs;

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Fontaine, RN, PhD, Principal Investigator — McGill University
Locations (12):
- Canada (12):
  - Anonyme L'Unite D'Intervention, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Indigenous Health Centre of Tiohtià:ke, Montreal, Quebec
  - L'Anonyme, Montreal, Quebec
  - Centre de réadaptation en dépendance de Québec (CRDQ), Québec, Quebec
  - Medicins du Monde, Montreal
  - Okanagan prison, Okanagan
  - SABSA Cooperative, Québec
  - Sioux Lookout First Nation Health Authority, Sioux Lookout
  - Ontario - Provincial correction, Toronto
  - Rapid Access Addiction Clinic St Paul's Hospital, Vancouver
  - Maamwesying North Shore Community Health Services, Wawa

IPD SHARING:
Plan to Share IPD: No
We won't share IPD, we will share aggregated and analyzed data.

REFERENCES:
- [Derived] Mooney M, Weight C, Biondi MJ, Grebely J, Kronfli N, Barnett T, Bruneau J, Dunn K, Elakpa DN, Etherington C, Greenaway C, Martel-Laferriere V, Mendlowitz A, Taylor N, Fontaine G. Scaling up point-of-care hepatitis C testing in Canada: protocol for a multilevel implementation science study of clinical processes, barriers, facilitators and implementation strategies (SCALE-POCT study). Implement Sci Commun. 2025 Dec 18. doi: 10.1186/s43058-025-00837-3. Online ahead of print. PMID 41408357